CLINICAL TRIAL: NCT02594930
Title: Comparison of Directed Versus Undirected Synovial Biopsy in Culture-negative Periprosthetic Joint Infections (With Preoperative Smears From the Skin) of the Knee and Evaluation of Outcome After Revision Joint Arthroplasty
Brief Title: Comparison of Two Different Techniques of Synovial Biopsy and Resistances of Cutaneous Smears in Suspected PPI
Acronym: COSPI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Technical University of Munich (Other)
Responsible Party: Principal Investigator, Harrasser, Dr., Technical University of Munich
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AAA-11/145
Record Dates: First submitted 2015-10-31; First posted 2015-11-03 (Estimated); Last update posted 2016-10-19 (Estimated); Status verified 2016-10

CONDITIONS: Infection of Total Knee Joint Prosthesis
Keywords: synovial biopsy; knee arthroplasty; infection
MeSH Terms: conditions — Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- undirected and directed biopsy (Experimental): Via an antero-lateral incision of the knee samples are taken without visual control; Afterwards an arthroscope is inserted and samples are taken from 5 defined regions of the knee (suprapatellar pouch, medial and lateral gutter, notch, Hoffa's fat pad)
  Interventions: Procedure: synovial biopsy of total knee arthroplasty

INTERVENTIONS:
Procedure: synovial biopsy of total knee arthroplasty — synovial biopsies are taken via two different techniques in the same patient to allow direct comparison of results

SUMMARY:
The purpose of this study is to determine whether an undirected synovial biopsy technique has the same accuracy in detecting periprosthetic joint infection in the knee as an arthroscopic assisted directed synovial biopsy technique.

DETAILED DESCRIPTION:
Successful treatment of an infected joint arthroplasty depends on correctly identifying the responsible pathogens. The value of a preoperative biopsy remains controversial. We compared the sensitivity and specificity of two techniques of synovial biopsy of knee joint arthroplasties suspicious for infection and asked whether the results correlate with intraoperative findings at revision.

ELIGIBILITY:
Inclusion Criteria:

* Chronic painful knee prosthesis planned for synovial biopsy to detect infection
* Culture-negative joint aspiration

Exclusion Criteria:

* Co-morbidities: Tumour disease, immune suppression

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-09; Primary Completion 2017-09 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
Correlation of microbiological and histological results of undirected and directed synovial biopsies | within the first 14 days after surgery
  5 microbiological samples and 1 histological sample are taken form the knee undirected via an antero-lateral approach. Afterwards the same sample numbers are taken under arthroscopic view. Correlation of results between those two methods are investigated. If infection is detected two-stage exchange of prosthesis is performed. At this surgery samples from synovia and the implant-bone interface are again taken and again investigated for correlation.

SECONDARY OUTCOMES:
Correlation of microbiological results from synovial biopsy with intraoperative findings at revision | within the first 14 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Ruediger Eisenhart-Rothe, Prof., Study Chair — Klinikum rechts der Isar, TU Munich
Locations (1):
- Klinikum rechts der Isar, Munich, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Scheele C, Krauel I, Pohlig F, Muehlhofer H, Gerdesmeyer L, Lasic I, Prodinger PM, Banke I, von Eisenhart-Rothe R, Harrasser N. Guided and Unguided Biopsy in the Diagnostic of Periprosthetic Infections of the Knee - Evaluation of an Evidence-based Algorithm. Z Orthop Unfall. 2019 Dec;157(6):684-694. doi: 10.1055/a-1034-0923. Epub 2019 Oct 28. English, German. PMID 31658475